CLINICAL TRIAL: NCT05738954
Title: Pattern Recognition and Anomaly Detection in Fetal Morphology Using Deep Learning and Statistical Learning
Acronym: PARADISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Craiova (Other)
Responsible Party: Sponsor
Other Study IDs: PARADISE
Record Dates: First submitted 2023-02-01; First posted 2023-02-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Congenital Abnormalities
Keywords: ultrasound; fetal morphology; view planes; deep learning; learning curves
MeSH Terms: conditions — Congenital Abnormalities | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Second trimester: Second trimester fetal morphology Collect patient data, anonymize and label it. Written informed consent or verbal recorded consent (if the participant lacks the ability to write or sign) will be obtained before performing the MS. In the unlikely event that some of the participants will withdraw their consent after the ultrasound has been performed, the data collected will not be used in the project. Data for publications and dataset will be previously made anonymous following standard practices. The participants will sign a GDPR form.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Collect patient data, anonymize and label it. Written informed consent or verbal recorded consent (if the participant lacks the ability to write or sign) will be obtained before performing the MS. In the unlikely event that some of the participants will withdraw their consent after the ultrasound has been performed, the data collected will not be used in the project. Data for publications and dataset will be previously made anonymous following standard practices. The participants will sign a GDPR form.
  The DL/SL algorithms will work in a competitive/collaborative way. Following the 'no-free-lunch' theorem, we shall use the competitive phase to establish the most suitable DL/SL technique for the identification and anomaly detection of each organ, and the collaborative phase to make all the algorithms work together in providing a 'second' opinion.

SUMMARY:
Congenital anomalies (CA) are the most encountered cause of fetal death, infant mortality and morbidity.7.9 million infants are born with CA yearly. Early detection of CA facilitates life-saving treatments and stops the progression of disabilities. CA can be diagnosed prenatally through Morphology Scan (MS). Discrepancies between pre and postnatal diagnosis of CA reach 29%. A correct interpretation of MS allows a detailed discussion regarding the prognosis with parents. The central feature of PARADISE is the development of a specialized intelligent system that embeds a committee of Deep Learning and Statistical Learning methods, which work together in a competitive/collaborative way to increase the performance of MS examinations by signaling CA. Using preclinical testing and clinical validation, the main goal will be the direct implementation into clinical practice. This multi-disciplinary project offers a unique integration of approaches, competences, breakthroughs in key applications in human, psychological, technological, and economical interest such as the 'smarter' healthcare system, opening new fields of research. PARADISE creates an environment that contributes significantly to the healthcare system, medical and pharma industries, scientific community, economy and ultimately to each individual. Its outcome will increase impact on the management of CA by enabling the establishment of detailed plans before birth, which will decrease morbidity and mortality in infants.

DETAILED DESCRIPTION:
Probe guidance: The IS guides the sonographer's probe for better acquisition of the fetal biometric plane - Basic scanning to be performed by non-expert(> 90% accuracy (AC)) Fetal biometric plane finder: The fetal planes are automatically detected, measured and stored - Insurance that all anatomical parts are checked (100% AC) Anomaly detection: unusual findings are signaled - Assistance in decision making (>90% AC)

ELIGIBILITY:
Inclusion Criteria:

* Second trimester pregnant women

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The pregnant women that have their second trimester morphology scan scheduled. They are included in the study consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Signal congenital anomalies | 32 months
  Number of congetinal anomalies found in a fetus at the second trimester morphology scan

CONTACTS AND LOCATIONS:
Overall Officials: Smaranda Belciug, Assoc. Prof., Principal Investigator — University of Craiova
Locations (1):
- University Emergency County Hospital, Craiova, Dolj, Romania

IPD SHARING:
Plan to Share IPD: Yes
Element 1: Data Type Primary and secondary data from RGB 2D ultrasound images (4000 images)
  The data can be used by researchers to further improve the diagnostic of congenital anomalies.
  Element 2: Related Tools, Software and/or Code:
  There will be no specific tools for accessing data.
  Element 4: Data Preservation, Access, and Associated Timelines
  A. Repository where scientific data and metadata will be archived:
  www.zenodo.org
  When and how long the scientific data will be made available:
  December 2024-December 2034
  Element 5: Access, Distribution, or Reuse Considerations Informed consent, anonymized data, privacy constraints and applicable ethical norms, national laws, privacy policies
  Element 6: Oversight of Data Management and Sharing:
  Renato Constantin Ivanescu- anonymizing the data and collecting it Dominic Iliescu, Rodica Nagy, Anca Ofiteru, Cristina Comanescu - gathering data Smaranda Belciug - overall supervision role for data management
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available in December 2024 and will be available until December 2034
Access Criteria: No criteria

REFERENCES:
- [Result] Belciug S. Learning deep neural networks' architectures using differential evolution. Case study: Medical imaging processing. Comput Biol Med. 2022 Jul;146:105623. doi: 10.1016/j.compbiomed.2022.105623. Epub 2022 May 17. PMID 35751202
- [Result] Belciug S, Ivanescu RC, Popa SD, Iliescu DG. Doctor/Data Scientist/Artificial Intelligence Communication Model. Case Study. Procedia Comput Sci. 2022;214:18-25. doi: 10.1016/j.procs.2022.11.143. Epub 2022 Dec 8. PMID 36514710
- [Derived] Belciug S. Autonomous fetal morphology scan: deep learning + clustering merger - the second pair of eyes behind the doctor. BMC Med Inform Decis Mak. 2024 Apr 19;24(1):102. doi: 10.1186/s12911-024-02505-3. PMID 38641580
- [Derived] Belciug S, Ivanescu RC, Serbanescu MS, Ispas F, Nagy R, Comanescu CM, Istrate-Ofiteru A, Iliescu DG. Pattern Recognition and Anomaly Detection in fetal morphology using Deep Learning and Statistical learning (PARADISE): protocol for the development of an intelligent decision support system using fetal morphology ultrasound scan to detect fetal congenital anomaly detection. BMJ Open. 2024 Feb 15;14(2):e077366. doi: 10.1136/bmjopen-2023-077366. PMID 38365300
- See also: Project website — https://www.paradise-pce.ro/